CLINICAL TRIAL: NCT00958555
Title: A Study of Predictive and Prognostic Markers in Patients With Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: NS02/04/09
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
1. To establish a retrospective compilation of clinical, histopathological, treatment and follow-up (clinic pathological) data of previous non-small cell lung cancer (NSCLC) cases.
2. To establish a prospective collection of clinic pathological information from NSCLC patients with corresponding blood and tissue samples
3. To discover and validate molecular biomarkers of survival and treatment outcome in NSCLC

One of the current difficulties in the management of lung cancer is the decision to treat and the type of treatment to select. Thus there is a need for additional prognostic (indicative of disease aggressiveness) and predictive (indicative of likely response to treatment) markers for lung cancer. To conduct a successful prognostic and predictive marker program, several factors are required, including: a comprehensive database linking clinical, histopathological, treatment and outcome characteristics of each case, a collection of samples linked to the database that is suitable for the testing of candidate markers, and a multi-disciplinary, interdepartmental level of expertise in the management of lung cancer.

Objective 1:

A review of the case records will be conducted to extract clinical, treatment and follow-up data

Objective 2:

Patients aged 21 years or more with newly diagnosed, untreated non-small cell lung cancer shall be approached for consent. Patients will be identified through the pathology records, and from the study investigators' clinic. After subject consent, baseline characteristics will be obtained. Follow up data on therapies received and toxicities encountered will be obtained. Tumor samples will be obtained only from patients with NSCLC undergoing surgery as part of routine clinical care. The surgical specimen will be sent to Pathology to verify the adequacy of the diagnostic sample as per usual practice. Blood will be collected at the baseline (or prior to any anti-cancer treatment) and will be sampled again at the time of relapse or disease progression. Collection will entail drawing 7ml blood into a Vacutainer CPT tube (Becton Dickinson, USA), centrifugation, extraction of a separated layer of mononuclear cells (MNC), labeling followed by storage below -80oC. The frequency of blood drawn will be about 1-5 times (7-35mls total). The number of times depends on whether the lung cancer relapses and in the advanced stage, how often the lung cancer relapses after treatment. DNA and RNA will be extracted by CSIS and stored in freezer space there. Stored samples will be used for investigation of prognostic and predictive markers of outcome and for discovery of novel molecular alterations

Objective 3:

Biomarker analysis of tumor and blood. Blood will be enriched for circulating tumor cells (CTC) using previously optimized methods (11) and DNA will be extracted from CTC and tumor using the Tri-Reagent (Molecular Research Center, Cincinatti, OH). DNA will be extracted from tumor, CTC and mononucleated cells and tested for somatic lung mutations by sequencing (2). Germline DNA will be analysed for genes linked to genetic risk for NSCLC and, for treatment toxicities, for genes related to NSCLC chemotherapy metabolic pathways.

Tissue microarray (TMA) is a high-throughput method of analysing large numbers of formalin-fixed, paraffin-embedded tumor at a minimal cost and effort. To analyse the expression of proteins of putative relevance to EGFR function, cell proliferation, angiogenesis, apoptosis, metastasis, and hormonal, TMA will be utilised. PTEN and C/EBPa will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed non-small cell lung cancer
* age 21 years or more
* untreated
* for the retrospective review, patients with a diagnosis of non-small cell lung cancer aged above 21 years or more

Exclusion Criteria:

* no consent
* if, in the investigator's opinion, the patient is unable to comply with study protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators for this protocol are clinicians and scientists in the departments of Cardiac/Thoracic and Vascular Surgery, Haematology and Oncology, Pathology, Radiation Oncology, Respiratory Medicine, and the Cancer Sciences Institute of Singapore (CSIS) from NUH, and NUS with major roles in their departments in the clinical management and/or research of lung cancer. Each will be providing access to clinical information and assisting in the collection and processing of samples, according to their resources and expertise.
Sampling Method: Probability Sample
Dates: Start 2009-04; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Sequist LV, Bell DW, Lynch TJ, Haber DA. Molecular predictors of response to epidermal growth factor receptor antagonists in non-small-cell lung cancer. J Clin Oncol. 2007 Feb 10;25(5):587-95. doi: 10.1200/JCO.2006.07.3585. PMID 17290067